CLINICAL TRIAL: NCT02316730
Title: Single-dose, Open, Randomized, Two-period, Crossover Comparative Bioavailability Study of Sanchi-Tongshu Capsule and Sanchi-Tongshu Capsule (Enteric Coated Pellets) in Chinese Healthy Adult Male Subjects
Brief Title: A Bioequivalence Study of Sanchi-Tongshu Capsule (Enteric Coated Pellets)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Factory of Chengdu HuaSun Group Inc., Ltd. (Industry)
Collaborators: West China Second University Hospital (Other); Sichuan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SQTS1212; ChiCTR-TTRCC-13003277 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2014-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sanchi-Tongshu Capsule (Enteric coated pellets) (Experimental): Sanchi-Tongshu Capsule (Enteric coated pellets) is developed by pharmaceutical factory of Chengdu Huasun Group Inc., 0.35g/capsule, containing 100mg of panaxatriol saponins (PTS).
  Interventions: Drug: Sanchi-Tongshu Capsule (Enteric coated pellets)
- Sanchi-Tongshu Capsule (Active Comparator): Sanchi-Tongshu Capsule is developed by pharmaceutical factory of Chengdu Huasun Group Inc., 0.2g/capsule, containing 100mg of panaxatriol saponins (PTS).
  Interventions: Drug: Sanchi-Tongshu Capsule

INTERVENTIONS:
Drug: Sanchi-Tongshu Capsule (Enteric coated pellets) — Take 0.7g (2 Capsules) of test preparation orally.
  Arms: Sanchi-Tongshu Capsule (Enteric coated pellets)
Drug: Sanchi-Tongshu Capsule — Take 0.4g (2 Capsules) of reference preparation orally.
  Arms: Sanchi-Tongshu Capsule

SUMMARY:
24 healthy male volunteers are to be assigned to take orally Sanchi-Tongshu Capsule (Enteric coated pellets) and Sanchi-Tongshu Capsule in fasting condition according to a randomized, crossover, self-control method, with ginsenoside Rg1, ginsenoside Re and notoginsenoside R1 as detection indicators. Establish the "blood drug concentration-time " curve, compare the bioequivalence of the main effective ingredients of the two preparations during the absorption process in human.

ELIGIBILITY:
Inclusion Criteria:

* The healthy male volunteers aged 18-40 years old;
* The body mass index is within 19-24, and the body weight is not less than 50kg( body mass index=body weight (kg)/height (M)2);
* All the examination indicators such as heart, liver, kidney, blood and so on are within normal range;
* The subjects should be without the addiction to smoking or alcohol, without drug abuse history and agree not to drink beverages containing caffeine during the trial;
* The subjects fully understand the objective, method and content of the trial, as well as the test preparation and reference preparation, and are willing to sign informed consent.

Exclusion Criteria:

* The subjects that are found to have any significant clinical diseases by direct questioning and comprehensive physical examination and laboratory examination before study;
* Allergic constitution, such as the patients with allergy history to two or more food and drugs; or those known to be allergic to the ingredient of the drug.
* The individuals with low possibility of enrollment (such as physically weak and so on) according to investigator's judgement;
* The patients that have any reasons considered by the investigator to prevent the subjects from finishing the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to 33 hours post dose(AUC0-33h) | Up to 33 hours post dose
Area under the plasma concentration-time curve from zero to infinity post dose(AUC0-∞) | Up to 33 hours post dose
Maximum observed concentration (Cmax ) | Up to 33 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Xihong Li, MD, Principal Investigator — West China Second University Hospital
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China